CLINICAL TRIAL: NCT00194844
Title: Caring Interventions for Couples Who Have Miscarried
Brief Title: Couples Miscarriage Healing Project:Randomized Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Kristen M. Swanson, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 01-1206-G 02; 5R01NR005343-04 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Miscarriage; Grief; Pregnancy Loss
Keywords: caring; miscarriage; grief; couples; counseling
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Nurse Caring
  Interventions: Behavioral: Nurse Caring
- 2 (Experimental): Self Caring
  Interventions: Behavioral: Self Caring
- 3 (Experimental): Combined Caring
  Interventions: Behavioral: Combined Caring
- 4 (No Intervention): This group is not treated and serves as control.

INTERVENTIONS:
Behavioral: Nurse Caring — Nurse Caring: Couples receive three one hour counseling session with a nurse interventionist at approximately 1, 5 and 11 weeks after enrollment. Content for the intervention comes from Swanson's phenomenologically derived Meaning of Miscarriage Model. The process for the intervention is based on Swanson's Theory of Caring.
  Arms: 1
Behavioral: Self Caring — Self Caring: Couples receive a mailed videotape and workbook at approximately 1, 5 and 11 weeks after enrollment. Content for the intervention comes from Swanson's phenomenologically derived Meaning of Miscarriage Model. The process for the intervention is based on Swanson's Theory of Caring.
  Arms: 2
Behavioral: Combined Caring — Combined Caring: Couples receive one counseling session from a nurse interventionist at approximately one week after enrollment. Upon completion of the session the nurse will hand the couple a self-caring videotape and workbook. Couples will be mailed an additional videotape and workbook at approximately 5 and 11 weeks after enrollment. Content for the intervention comes from Swanson's phenomenologically derived Meaning of Miscarriage Model. The process for the intervention is based on Swanson's Theory of Caring.
  Arms: 3

SUMMARY:
This is a randomized trial of three caring based interventions to see if we can help couples heal after miscarriage. All three are based on Swanson's theory of caring and Meaning of Miscarriage Model. The first, nurse caring, consists of three counseling sessions with a nurse. The second intervention, self-caring, involves watching three videotapes and completing three workbooks. The third, combined caring, involves receiving one counseling session with a nurse followed up with the three videotapes and workbooks. There is also a control group that receives no intervention. All interventions are administered at 1, 6, and 11 weeks after study enrollment. Couples can enroll who are no more than 12 weeks post miscarriage of a pregnancy that ended at 20 weeks gestation or less. At 1, 6, 16, and 52 weeks post enrollment we ask couples to complete mailed booklets that contain a variety of research questionnaires about their emotional health, integration of loss, and couple relationship.

DETAILED DESCRIPTION:
The purpose of this randomized study is to compare the effects of nurse caring (3 nurse counseling sessions), self-caring (3 home-delivered videotapes and journals), combined caring (1 nurse counseling plus 3 videotapes and journals) and no intervention (control) on the emotional healing, integration of loss, and couple well-being of women and their partners (husbands or male mates) in the first year after miscarrying. A recent IoM [41] report claims one of the greatest obstacles to determining effectiveness of home-based interventions is getting clients to complete treatment protocols, thus the combined-caring group is included to determine if nurse endorsement of the videotape/journal modules enhances adherence and increases the efficacy of the self-caring protocol. All intervention materials are based on Swanson's middle-range caring theory [109,112] and Meaning of Miscarriage Model [116]. Both frameworks were phenomenologically derived and subsequently applied and tested in the Miscarriage Caring Project (MCP), a randomized trial of the effects of 3 caring-based nurse counseling sessions on women's emotional well-being and integration of loss in the first year after miscarriage [115]. The MCP is the only randomized post-miscarriage intervention that has led to significant positive mental health outcomes for women.

There are no published studies of interventions that have led to significant outcomes for men or couples post miscarriage. Yet, the PI's experience counseling couples groups (also based on the caring theory and miscarriage model) has provided consistent, albeit anecdotal, evidence that including partners helps couples to reach out to each other, integrate miscarriage into their lives, and resolve grieving. Therefore, this project focuses on women and their partners (spouses or male mates in a committed relationship). An additional goal is to determine if an innovative, easily delivered, low-cost video/journal intervention is as effective as interpersonal counseling in assisting women and their partners to emotionally heal, integrate loss, and experience couple well being in the first year after miscarriage.

The procedural aims are to:

1. Develop an empirically derived self-caring intervention for couples who have miscarried. This home-delivered intervention will be a series of three modules consisting of broadcast quality videotapes ("Miscarriage: Caring and Healing") and journal assignments. (drafts are in Appendices B.1 to B.3.)
2. Train nurses to deliver a three session caring-based counseling intervention to couples.
3. Randomly assign couples who recently miscarried to one of four groups: group I (nurse caring) will receive three counseling sessions. Couples in group II (combined-caring) will receive one counseling session plus three self-caring videotape / journal modules; Group III (self-caring) will receive the three self-caring videotape / journal modules. Group IV (control) will receive no intervention.

There are four hypothesis-testing specific aims and one exploratory research aim:

1. Compared to controls, women and their partners who receive nurse, combined, or self-caring will report significantly more emotional healing, stronger integration of loss, and greater couple well-being in the first year subsequent to miscarriage.
2. Comparing the three modes of delivering caring (nurse, combined, and self), for women and their partners, there will be no differences in emotional healing, integration of loss, and couple well-being
3. Comparing self-caring to combined-caring, for women and their partners, within and across intervention times, there will be no differences in intervention adherence and / or evaluation scores.
4. Comparing the nurse-caring group to the combined-caring group, for women and their partners, there will be no differences in ratings of counselor empathy and caring at the first counseling session.
5. Determine associations amongst background variables, intervention monitoring scores, intervening variables, emotional healing, integration of loss, and couple well-being for women and their partners at 1 week, 6 weeks, 4 months and 1 year post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. unexpected, unplanned loss of pregnancy prior to 20 weeks gestation
2. no more than 12 weeks post loss
3. both the woman who miscarried and her male mate agree to participate
4. able to read, write, and speak in English
5. If 18 or older in a self proclaimed committed heterosexual relationship
6. If married, may be under 18

Exclusion Criteria:

1. non heterosexual couples
2. not geographically accessible to the Puget Sound area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2001-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Nikcevic Miscarriage Grief Inventory | first year after miscarriage

SECONDARY OUTCOMES:
Depression(CES-D); Mood Disturbances(POMS); Coping (Modified Folkman and Lazarus Ways of Coping); Emotional Strength (Swanson); Impact of Miscarriage (Swanson) | first year after miscarriage
Couple relationship Mate Caring (Swanson); Support of Mate and Others (Brown); Intimacy (PAIR); Professional Caring (Swanson) | first year after miscarriage

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Swanson, RN, PhD, Principal Investigator — University of Washington School of Nursing
Locations (1):
- University of Washington School of Nursing, Seattle, Washington, United States